CLINICAL TRIAL: NCT06647563
Title: A Randomized Controlled Study of Toripalimab Combined With Chemotherapy or With Chemotherapy/Cetuximab as Neoadjuvant Therapy for Locally Advanced Squamous Cell Carcinoma of the Head and Neck (Neo-ICT)
Brief Title: Neoadjuvant Toripalimab + Chemotherapy ± Cetuximab in Locally Advanced Head and Neck Squamous Cell Carcinoma (Neo-ICT)
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Yue He, MD, M.D., Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JYKQ-2024-105
Record Dates: First submitted 2024-10-13; First posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
Keywords: Programmed Cell Death-1 (PD1, PD-1); Head and Neck Squamous Cell Carcinoma; Toripalimab; Albumin-bound paclitaxel; Carboplatin; Cetuximab; Neoadjuvant
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — toripalimab; spartalizumab; Cetuximab; Albumin-Bound Paclitaxel; Carboplatin; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Toripalimab + Chemotherapy + Cetuximab + SOC (Immunotherapy+ chemotherapy+targeted therapy, ICT) (Experimental): Participants will receive an intravenous (IV) infusion of Toripalimab 240mg on Day 1, Albumin-bound Paclitaxel 125mg/m^2 on Days 1 and 8, Carboplatin with an area under the curve (AUC) of 5 on Day 1, and Cetuximab 400mg/m^2 on Day 1, followed by Cetuximab 250mg/m^2 on Day 1 of each subsequent week. The treatment is given in 21-day cycles for a total of two cycles. Afterward, participants will proceed to the standard of care (SOC), which includes surgical intervention and postoperative radiotherapy. Following surgical resection, high-risk participants will receive standard radiotherapy plus Cisplatin 100 mg/m^2 via intravenous infusion on Day 1, every 3 weeks (Q3W) for three 21-day cycles. Low-risk participants will receive only standard radiotherapy. Subsequently, participants will receive Toripalimab 240mg every 21-day cycle for a total of 15 cycles.
  Interventions: Biological: Toripalimab; Biological: Cetuximab; Drug: Albumin-Bound Paclitaxel; Drug: Carboplatin; Drug: Cisplatin; Radiation: Radiotherapy 60 Gray/day; Radiation: Radiotherapy 66 Gray/day; Radiation: Radiotherapy 70 Gray/day
- Toripalimab + Chemotherapy + SOC (Immunotherapy+ chemotherapy, IC) (Experimental): Participants will receive an intravenous (IV) infusion of Toripalimab 240mg on Day 1, Albumin-bound Paclitaxel 125mg/m^2 on Days 1 and 8, Carboplatin with an area under the curve (AUC) of 5 on Day 1. The treatment is given in 21-day cycles for a total of two cycles. Afterward, participants will proceed to the standard of care (SOC), which includes surgical intervention and postoperative radiotherapy. Following surgical resection, high-risk participants will receive standard radiotherapy plus Cisplatin 100 mg/m^2 via intravenous infusion on Day 1, every 3 weeks (Q3W) for three 21-day cycles. Low-risk participants will receive only standard radiotherapy. Subsequently, participants will receive Toripalimab 240mg every 21-day cycle for a total of 15 cycles.
  Interventions: Biological: Toripalimab; Drug: Albumin-Bound Paclitaxel; Drug: Carboplatin; Drug: Cisplatin; Radiation: Radiotherapy 60 Gray/day; Radiation: Radiotherapy 66 Gray/day; Radiation: Radiotherapy 70 Gray/day
- No Neoadjuvant + SOC (Control) (Active Comparator): Participants will receive the standard of care (SOC) with no neoadjuvant prior to surgery. Following surgical resection, high-risk participants will receive standard radiotherapy plus Cisplatin 100 mg/m^2 via intravenous infusion on Day 1, every 3 weeks (Q3W) for three 21-day cycles. Low-risk participants will receive only standard radiotherapy.
  Interventions: Drug: Cisplatin; Radiation: Radiotherapy 60 Gray/day; Radiation: Radiotherapy 66 Gray/day; Radiation: Radiotherapy 70 Gray/day

INTERVENTIONS:
Biological: Toripalimab — Specified dose on specified days
  Other Names: PD-1 antibody
  Arms: Toripalimab + Chemotherapy + Cetuximab + SOC (Immunotherapy+ chemotherapy+targeted therapy, ICT); Toripalimab + Chemotherapy + SOC (Immunotherapy+ chemotherapy, IC)
Biological: Cetuximab — Specified dose on specified days
  Other Names: EGFR antibody
  Arms: Toripalimab + Chemotherapy + Cetuximab + SOC (Immunotherapy+ chemotherapy+targeted therapy, ICT)
Drug: Albumin-Bound Paclitaxel — Specified dose on specified days
  Arms: Toripalimab + Chemotherapy + Cetuximab + SOC (Immunotherapy+ chemotherapy+targeted therapy, ICT); Toripalimab + Chemotherapy + SOC (Immunotherapy+ chemotherapy, IC)
Drug: Carboplatin — Specified dose on specified days
  Arms: Toripalimab + Chemotherapy + Cetuximab + SOC (Immunotherapy+ chemotherapy+targeted therapy, ICT); Toripalimab + Chemotherapy + SOC (Immunotherapy+ chemotherapy, IC)
Drug: Cisplatin — Specified dose on specified days
Radiation: Radiotherapy 60 Gray/day — Low risk participants administered 2 Gray/day in 30 fractions. Administered using intensity modulated radiation therapy.
Radiation: Radiotherapy 66 Gray/day — High risk participants administered 2 Gray/day in 33 fractions. Administered using intensity modulated radiation therapy.
Radiation: Radiotherapy 70 Gray/day — Participants with gross residual disease administered 2 Gray/day in 35 fractions. Administered using intensity modulated radiation therapy.

SUMMARY:
This study is a randomized, active-controlled, open-label clinical trial for participants with newly diagnosed Stage III-IVb, resectable, locoregionally advanced head and neck squamous cell carcinoma (LA-HNSCC). The study consists of two experimental arms and one control arm. Participants in Experimental Arm A will receive two cycles of Toripalimab, albumin-bound paclitaxel, carboplatin, and cetuximab prior to surgery. Participants in Experimental Arm B will receive two cycles of Toripalimab, albumin-bound paclitaxel, and carboplatin before surgical intervention. Following the surgical procedure, individuals in both Experimental Arm A and B will continue to receive 15 cycles of Toripalimab. The Control Arm will undergo the current standard treatment without preoperative drug intervention. Postoperatively, participants will be administered postoperative radiotherapy or chemoradiotherapy based on their recurrence risk. The primary study hypotheses are that the treatments in the Experimental Arms will improve the 2-year event-free survival (EFS) rates compared to the standard control treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed squamous cell carcinoma of the head and neck (excluding nasopharyngeal cancer);
2. Male or female, aged 18-75 years;
3. Clinical stage III-IVb (AJCC 8th edition TNM stage) and operable patients; if oropharyngeal squamous cell carcinoma (P16-), the stage is III-IVb; if oropharyngeal squamous cell carcinoma (P16+), the stage is III;
4. No prior antitumor therapy including radiotherapy, chemotherapy, immunotherapy or biological therapy for the current tumor;
5. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1;
6. Life expectancy ≥ 6 months;
7. No obvious contraindications to immunotherapy, radiochemotherapy, or surgical treatment;
8. Willing to accept surgical treatment;
9. The level of main organ function meets the following criteria:

   1. Routine blood tests: WBC ≥ 4.0 × 10^9/L, ANC ≥ 1.5 × 10^9/L, PLT ≥ 100 × 10^9/L, Hb ≥ 90 g/L (no blood transfusion or blood products within 14 days, no correction with G-CSF and other hematopoietic growth factors);
   2. Biochemical assessments: serum albumin ≥ 3.0 g/dL (30 g/L), TBIL ≤ 1.5 × ULN, ALT, AST ≤ 2.5 × ULN, BUN and CRE ≤ 1.5 × ULN or creatinine clearance ≥ 60 mL/min (Cockcroft-Gault formula);
   3. Adequate coagulation function: defined as international normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 × ULN; If the subject is receiving anticoagulant therapy, PT should be within the proposed therapeutic range of the anticoagulant;
10. Women of childbearing potential must have a negative pregnancy test result (serum or urine), conducted within seven days prior to enrollment and agree to use effective contraception during the study period and for six months post last dose of anti-PD-1 antibody administration. Male subjects with female partners who are capable of conception must also utilize effective contraception throughout this study duration and for six months after their final dose anti-PD-1 antibody;
11. Willingness to participate in this study by signing an informed consent form, while exhibiting strong compliance and readiness to cooperate with follow-up procedures.

Exclusion Criteria:

1. Previous treatment with anti-PD-1/PD-L1 antibody, anti-PD-L2 antibody, anti-CD137 antibody, anti-CTLA-4 antibody, or other drugs/antibodies targeting T cell co-stimulation or checkpoint pathway;
2. Active autoimmune disease. Subjects in stable condition who do not require systemic immunosuppressive therapy are permitted; examples include type I diabetes mellitus, hypothyroidism requiring only hormone replacement therapy, and skin conditions that do not necessitate systemic treatment (e.g., vitiligo, psoriasis, alopecia).
3. Patients with congenital or acquired immunodeficiency (e.g., HIV infection), active hepatitis B (HBV-DNA ≥ 10^4 copies/ml) or hepatitis C (positive antibody for HCV, and HCV-RNA above the lower limit of detection of the analytical procedure);
4. Known allergy to the study drug or any of its excipients; or serious allergic reaction to other monoclonal antibodies.
5. The occurrence of any of the following conditions within 6 months prior to randomization: myocardial infarction, severe/unstable angina pectoris, NYHA class II or higher cardiac insufficiency, clinically significant supraventricular or ventricular arrhythmias, and symptomatic congestive heart failure.
6. Vaccination with live vaccines within 4 weeks prior to the first dose of the study drug. Inactivated virus vaccine can be administered for seasonal flu, but not attenuated live influenza vaccines administered intranasally.
7. Known history of allogeneic organ transplant or allogeneic stem cell transplant.
8. The history of drug addiction and the abuse of psychoactive substances.
9. Pregnant or breastfeeding women.
10. Any other malignant neoplasm diagnosed within 5 years prior to study entry, except for carcinoma that is amenable to local treatment and has been cured, such as basal cell carcinoma or squamous cell carcinoma of the skin, superficial bladder cancer, cervical carcinoma in situ, carcinoma in situ of breast ductal, and papillary thyroid cancer.
11. Patients with other significant physical or mental health conditions, or laboratory test abnormalities that may elevate the risk of participation in the study or compromise the integrity of the study results, as determined by the investigators, are deemed unsuitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 355 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2029-09-30 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
ICT vs Control: Two-Year Event-free Survival (EFS) rate | Up to ~72 months
  Two-Year Event-free Survival (EFS) rate defined as the proportion of participants who have not experienced any EFS events by the 2-year mark from randomization, out of all participants in the arm.
  EFS events: any progression of disease precluding surgery, progression or recurrence disease after surgery, death due to any cause, or occurrence of a second primary tumor. Participants who don't undergo surgery for reason other than progression will be considered to have an event at progression or death.
  EFS: The time from randomization, until the first documented occurrence of EFS event.
  Per protocol, Two-Year EFS rate in the ICT arm will be compared to the control arm as a pre-specified primary analysis of the Intent-To-Treat (ITT) population.
IC vs Control: Two-Year EFS rate | Up to ~72 months
  Two-Year EFS rate defined as the proportion of participants who have not experienced any EFS events by the 2-year mark from randomization, out of all participants in the arm.
  EFS events: any progression of disease precluding surgery, progression or recurrence disease after surgery, death due to any cause, or occurrence of a second primary tumor. Participants who don't undergo surgery for reason other than progression will be considered to have an event at progression or death.
  EFS: The time from randomization, until the first documented occurrence of EFS event.
  Per protocol, Two-Year EFS rate in the IC arm will be compared to the control arm as a pre-specified primary analysis of the Intent-To-Treat (ITT) population.

SECONDARY OUTCOMES:
ICT vs Control: Overall Survival (OS) | Up to ~96 months
  OS is the time from randomization to death due to any cause. Per protocol, OS in the ICT arm will be compared to the control arm as a pre-specified secondary analysis of the ITT population.
IC vs Control: OS | Up to ~96 months
  OS is the time from randomization to death due to any cause. Per protocol, OS in the IC arm will be compared to the control arm as a pre-specified secondary analysis of the ITT population.
ICT vs IC: Major Pathological Response (MPR) | Up to ~40 months
  The percentage of participants with a major pathological response (MPR) as assessed by the Central Pathologist at the time of definitive surgery. MPR is defined as ≤10% invasive squamous cell carcinoma within the resected primary tumor specimen and all the sampled regional lymph nodes.
  Per protocol, MPR in the ICT arm will be compared to the IC arm as a pre-specified secondary analysis of the ITT population.
ICT vs IC: Pathological Complete Response (PCR) | Up to ~40 months
  he percentage of participants with a pathological complete response (PCR) as assessed by the central pathologist at the time of definitive surgery. PCR is defined as having no residual invasive squamous cell carcinoma within the resected primary tumor specimen and all sampled regional lymph nodes.
  Per protocol, PCR in the ICT arm will be compared to the IC arm as a pre-specified secondary analysis of the ITT population.
ICT vs IC: Objective Response Rate (ORR) | Up to ~40 months
  According to Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), Objective Response Rate (ORR) assesses the proportion of subjects with complete response (CR) and partial response (PR).
  Per RECIST v1.1 criteria for target lesions and assessed by MRI or CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Per protocol, ORR in the ICT arm will be compared to the IC arm as a pre-specified secondary analysis of the ITT population.
ICT vs Control: Three-Year EFS rate | Up to ~84 months
  Three-Year EFS rate defined as the proportion of participants who have not experienced any EFS events by the 3-year mark from randomization, out of all participants in the arm.
  EFS events: any progression of disease precluding surgery, progression or recurrence disease after surgery, death due to any cause, or occurrence of a second primary tumor. Participants who don't undergo surgery for reason other than progression will be considered to have an event at progression or death.
  EFS: The time from randomization, until the first documented occurrence of EFS event.
  Per protocol, Three-Year EFS rate in the ICT arm will be compared to the control arm as a pre-specified secondary analysis of the ITT population.
ICT vs Control: Five-Year EFS rate | Up to ~96 months
  Five-Year EFS rate defined as the proportion of participants who have not experienced any EFS events by the 5-year mark from randomization, out of all participants in the arm.
  EFS events: any progression of disease precluding surgery, progression or recurrence disease after surgery, death due to any cause, or occurrence of a second primary tumor. Participants who don't undergo surgery for reason other than progression will be considered to have an event at progression or death.
  EFS: The time from randomization, until the first documented occurrence of EFS event.
  Per protocol, Five-Year EFS rate in the ICT arm will be compared to the control arm as a pre-specified secondary analysis of the ITT population.
IC vs Control: Three-Year EFS rate | Up to ~84 months
  Three-Year EFS rate defined as the proportion of participants who have not experienced any EFS events by the 3-year mark from randomization, out of all participants in the arm.
  EFS events: any progression of disease precluding surgery, progression or recurrence disease after surgery, death due to any cause, or occurrence of a second primary tumor. Participants who don't undergo surgery for reason other than progression will be considered to have an event at progression or death.
  EFS: The time from randomization, until the first documented occurrence of EFS event.
  Per protocol, Three-Year EFS rate in the IC arm will be compared to the control arm as a pre-specified secondary analysis of the ITT population.
IC vs Control: Five-Year EFS rate | Up to ~96 months
  Five-Year EFS rate defined as the proportion of participants who have not experienced any EFS events by the 5-year mark from randomization, out of all participants in the arm.
  EFS events: any progression of disease precluding surgery, progression or recurrence disease after surgery, death due to any cause, or occurrence of a second primary tumor. Participants who don't undergo surgery for reason other than progression will be considered to have an event at progression or death.
  EFS: The time from randomization, until the first documented occurrence of EFS event.
  Per protocol, Five-Year EFS rate in the IC arm will be compared to the control arm as a pre-specified secondary analysis of the ITT population.
ICT vs IC: Two-Year EFS rate | Up to ~72 months
  Two-Year EFS rate defined as the proportion of participants who have not experienced any EFS events by the 2-year mark from randomization, out of all participants in the arm.
  EFS events: any progression of disease precluding surgery, progression or recurrence disease after surgery, death due to any cause, or occurrence of a second primary tumor. Participants who don't undergo surgery for reason other than progression will be considered to have an event at progression or death.
  EFS: The time from randomization, until the first documented occurrence of EFS event.
  Per protocol, Two-Year EFS rate in the ICT arm will be compared to the IC arm as a pre-specified secondary analysis of the ITT population.
ICT vs IC: Three-Year EFS rate | Up to ~84 months
  Three-Year EFS rate defined as the proportion of participants who have not experienced any EFS events by the 3-year mark from randomization, out of all participants in the arm.
  EFS events: any progression of disease precluding surgery, progression or recurrence disease after surgery, death due to any cause, or occurrence of a second primary tumor. Participants who don't undergo surgery for reason other than progression will be considered to have an event at progression or death.
  EFS: The time from randomization, until the first documented occurrence of EFS event.
  Per protocol, Three-Year EFS rate in the ICT arm will be compared to the IC arm as a pre-specified secondary analysis of the ITT population.
ICT vs IC: Five-Year EFS rate | Up to ~96 months
  Five-Year EFS rate defined as the proportion of participants who have not experienced any EFS events by the 5-year mark from randomization, out of all participants in the arm.
  EFS events: any progression of disease precluding surgery, progression or recurrence disease after surgery, death due to any cause, or occurrence of a second primary tumor. Participants who don't undergo surgery for reason other than progression will be considered to have an event at progression or death.
  EFS: The time from randomization, until the first documented occurrence of EFS event.
  Per protocol, Five-Year EFS rate in the ICT arm will be compared to the IC arm as a pre-specified secondary analysis of the ITT population.
ICT vs IC vs Control: Locoregional recurrence-free survival (LRFS) rate | Up to ~96 months
  The Two-Year, Three-Year, and Five-Year LRFS rates refer to the proportions of participants who have not experienced locoregional recurrence and are still alive at 2, 3, and 5 years post-randomization, respectively, out of all participants in the arm.
  Per protocol, the LRFS rate will be compared between the ICT, IC, and Control arms.
ICT vs IC vs Control: Distant Disease-free Survival (DDFS) rate | Up to ~96 months
  Two-Year, Three-Year, and Five-Year DDFS rates refer to the proportion of patients who have not experienced distant metastasis and are still alive at 2, 3, and 5 years post-randomization, out of all participants in the arm.
  Per protocol, the DDFS rate will be compared between the ICT, IC, and Control arms.
ICT vs IC vs Control: Change From Baseline in Global Health Status/Quality of Life Scale (GHS/QoL) | Up to ~96 months
  Change from baseline in the combined score of global health status (GHS)/quality of life (QoL) using the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Core Questionnaire (EORTC QLQ-C30) items 29 and 30. Participant responses to questions regarding overall health/QoL will be scored on a 7-point scale (1=Very poor to 7=Excellent) with a higher score indicating better overall health status.
ICT vs IC vs Control: Change From Baseline in Global Health Status/Physical Functioning Scales | Up to ~96 months
  Change from baseline in the combined score of physical functioning scale using the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Core Questionnaire (EORTC QLQ-C30) items 1 through 5. Participant responses to questions regarding their physical functioning will be scored on a 4-point scale (1=Not at All to 4=Very Much) with a higher score indicating worse physical functioning.
ICT vs IC vs Control: Change from Baseline in Swallowing, Speech, and Pain Symptoms | Up to ~96 months
  Change from baseline in the combined score of swallowing, speech, and pain symptoms using the European Organization for Research and Treatment of Cancer Head and Neck Questionnaire (EORTC QLQ-H&N35) items 31-38, 46, and 53-54. Participant responses to questions regarding problems with swallowing, speech and pain in the mouth will be scored on a 4-point scale (1=Not at all to 4=Very much) with a higher score indicating more problems.
ICT vs IC vs Control: Percentage of Participants Experiencing An Adverse Event (AEs) | Up to ~96 months
  Percentage of participants experiencing any sign, symptom, disease, or worsening of preexisting condition temporally associated with study therapy and irrespective of causality to study therapy.
ICT vs IC: Percentage of Participants Discontinuing Study Drug Due to AEs | Up to ~48 months
  Percentage of participants discontinuing study drug due to an AE.
ICT vs IC: OS | Up to ~96 months
  OS is the time from randomization to death due to any cause. Per protocol, OS in the ICT arm will be compared to the IC arm as a pre-specified secondary analysis of the ITT population.

CONTACTS AND LOCATIONS:
Overall Officials: Yue He, M.D., Principal Investigator — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University School of Medicine

IPD SHARING:
Plan to Share IPD: No